CLINICAL TRIAL: NCT04887142
Title: Biochemical, Inflammatory and Genetic Factors in Patients With COVID-19
Brief Title: Predictors of Disease Severity in COVID-19 Patients
Acronym: VIRIONUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zeljko Mijailovic (Other)
Responsible Party: Sponsor-Investigator, Zeljko Mijailovic, Principal Investigator, University of Kragujevac
Organization: University of Kragujevac (Other)
Other Study IDs: 01/20-405
Record Dates: First submitted 2021-05-08; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: COVID-19; Inpatients; Risk Factors; Treatment Outcome; Observational Study
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimen, serum, white cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The discharged subjects: The COVID-19 inpatients treated with standard care who survived the disease and discharged from hospital.
  Interventions: Other: Standard of health care
- The deceased subjects: The COVID-19 inpatients treated with standard care who died from the disease.
  Interventions: Other: Standard of health care

INTERVENTIONS:
Other: Standard of health care — The patients in this observational study will be exposed to the standard health care interventions according to the hospital diagnostic and treatment protocols and procedures and clinical judgment of the treating physicians.

SUMMARY:
The primary goal of the VIRIONUM project is to analyze the association of clinical, socio-demographic characteristics of patients and their genetic polymorphism, inflammatory and other biochemical markers with disease progression and death in subjects with COVID-19 disease. The research is an observational, cohort study with nested-case control design, including adult, male and female COVID-19 inpatients. Primary dependent variable will be outcome of disease, defined as discharge from the hospital or death. The outcomes and putative risk factors will be analyzed using binary logistic regressions. The proposed multi- and inter-disciplinary study should provide additional scientific evidence about risk factors for the development of severe forms of the disease and the COVID-19-related death.

DETAILED DESCRIPTION:
Background: Severe acute respiratory syndrome 2 (SARS-CoV-2) is etiological agent of heterogeneous corona-virus disease 19 (COVID-19), which clinical condition range from asymptomatic or mild to critically severe with high odds for fatal outcome. Since the pathophysiological pathways of COVID-19 disease development are not fully elucidated, resulting in repeated changes in treatment plans, there is an unmet need for more research into genetic, biochemical, immunological, and clinical predictive indicators of better outcomes in COVID-19 patients.

Aim: The VIRIONUM project's main aim is to investigate the relation between genetic polymorphisms, inflammatory and other biochemical markers, and disease severity and mortality in COVID-19-infected hospitalized patients.

Method and patients: The observational nested case-control clinical study will be conducted in at least 1019 COVID-19 patients. The genetic polymorphisms (ACE2, IFNL3/4 and TMPRSS2), serum concentration of soluble ACE2 and the pro- and anti-inflammatory cytokines, blood concentration of common inflammatory and other biomarkers, peripheral blood mononuclear leukocyte (PBMC) phenotype, demographic and clinical risk factors will be monitored as independent variables, while the dependent variables will be the outcome of the disease and the severity of the clinical condition. Genotyping will be performed by Real-Time PCR method, and serum concentrations of ACE2 and pro- and anti-inflammatory cytokines by ELISA method, and PBMC phenotype by flow cytometry. The disease severity will be assessed according to WHO criteria.

Expected results: The findings of this clinical study will contribute to understanding of significant genetic, biochemical, and clinical determinants of severity and lethal outcomes in COVID-19 patients, as well as, creation of set of recommendations for individuals at higher risk - future, evidence-based, targeted and individualized approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult age, 18 years old or more
* Male or female
* Hospitalization for COVID-19 after confirmation by SARS-CoV-2 rapid antigen test or RT-PCR
* Voluntary written consent of the subject to participate

Exclusion Criteria:

* Pregnant and breastfeeding women
* Fatal outcome during the first 24 hours of hospitalization
* Inability to collect the necessary study data
* Declining of the subject to voluntary participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of both sexes with different socio-demographic and clinical characteristics, who were hospitalized due to COVID-19. The decision on hospitalization and further treatment of patients is at the discretion of the attending physicians. All participants will be prospectively followed during their hospital stay. Patients will be included in the study if they are at least 18 years old and if they give voluntary written consent to participate. Pregnant and breastfeeding women, patients transferred from other hospitals and those who die during the first 24 hours of hospitalization will be excluded. In this study, stratification of participants according to age to those older than 65 years and younger is provided only for the purposes of statistical data processing and analyse.
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Fatal Outcome | Up to 6 weeks from recruitment to hospital discharge or death
  Case fatality ratio will be calculated as the proportion of patients who died from all causes (all-cause mortality) compared to the total number of patients

SECONDARY OUTCOMES:
Ordinal Scale for Clinical Improvement | Up to 6 weeks from recruitment to hospital discharge or death
  Patients' COVID-19 severity and clinical improvement will be assessed according to the recommendations of World Health Organization using Ordinal Scale for Clinical Improvement and the patient state will be classified as mild (score 4 or less) or severe (score 5 or more).

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Baskic, MD PHD, Study Chair — Faculty of Medical Sciences
Locations (5):
- Spitali Amerikan, Tirana, Albania
- General Hospital "Prim. dr. Abdulah Nakaš", Sarajevo, Bosnia and Herzegovina
- KBC Rijeka, University of Rijeka, Rijeka, Croatia
- University of Montenegro, Faculty of Medicine, Podgorica, Montenegro
- Faculty of Medical Sciences, University Clinical Center Kragujevac, Kragujevac, Srbija, Serbia

IPD SHARING:
Plan to Share IPD: No